CLINICAL TRIAL: NCT01625702
Title: Clinical Significance of Circulating Tumor Cells (CTCs) in Blood of Patients With Advanced/Metastatic Gastric Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Director of GI oncology, Peking University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CGOG5001
Record Dates: First submitted 2012-06-13; First posted 2012-06-21 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Gastric Cancer
Keywords: no-prior chemotherapy
MeSH Terms: conditions — Stomach Neoplasms

ARMS (2):
- cisplatin plus capecitabine (Experimental): gastric cancer patients treated with capecitabine/cisplatin
  Interventions: Device: CellSearch® CTC kit
- capecitabine plus paclitaxel (Experimental): gastric cancer patients treated with capecitabine/paclitaxel
  Interventions: Device: CellSearch® CTC kit

INTERVENTIONS:
Device: CellSearch® CTC kit — Collect peripheral blood sample of 100 gastric cancer patients pre-chemotherapy treated with capecitabine/paclitaxel (XPa) and capecitabine/cisplatin (XP) and post two cycles of chemotherapy(response evaluation).
  Blood samples will be transferred to central lab to detect CTCs by Cellsearch kit.
  Tumor response evaluation will be performed after two cycles of chemotherapy by CT/MRI based on RECIST. Clinical data, including tumor stage, metastastic organ, chemotherapy regimen, objective response, progression free survival, overall survival, etc, will be collected according to study protocol.

SUMMARY:
To identify the correlation of CTCs with clinical prognosis in advanced/metastatic gastric cancer. Confirm the presence of CTCs are sensitive for monitoring response to chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Having signed informed consent
* Age≥ 18 years old
* Histologically confirmed gastric adenocarcinoma
* Unresectable recurrent or metastatic disease
* Previous neo-adjuvant or adjuvant treatment for gastric cancer, if applicable, more than 6 months
* Previous chemotherapy with capecitabine or cisplatin, if applicable, more than 12 months.
* Measurable disease according to the RECIST criteria
* Karnofsky performance status ≥60
* Life expectancy of ≥2 month
* No prior radiotherapy except radiotherapy at non-target lesion of the study more than 4 weeks
* ALT and AST<2.5 times ULN (≤5 times ULN in patients with liver metastases)
* Serum albumin level ≥3.0g/dL
* Serum AKP < 2.5 times ULN
* Serum creatinine <ULN, and CCr < 60ml/min
* Bilirubin level < 1.5 ULN
* WBC>3,000/mm3, absolute neutrophil count ≥2000/mm3, platelet>100,000/mm3, Hb>9g/dl

Exclusion Criteria:

* Brain metastasis (known or suspected)
* Previous systemic therapy for metastatic gastric cancer
* Inability to take oral medication
* Previous therapy targeting at angiogenesis or vasculogenesis pathway or other targeted therapy
* Surgery (excluding diagnostic biopsy) within 4 weeks prior to study entry Contraindications of nuclear magnetic resonance image such as fitment of cardiac pacemaker , nerve stimulator, or aneurysm clip, and metallic foreign body in eye ball and so on.
* Allergic constitution or allergic history to protium biologic product or any investigating agents.
* Severe heart disease or such history as recorded congestive heart failure, uncontrolled cardiac arrhythmia, angina pectoris needing medication, cardiac valve disease, severe abnormal ECG findings, cardiac infarction , or retractable hypertension.
* Pregnancy or lactation period
* Any investigational agent within the past 28 days
* Other previous malignancy within 5 year, except non-melanoma skin cancer
* Previous adjuvant therapy with capecitabine+platinum,
* Pre-existing neuropathy>grade 1
* Legal incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2012-06; Primary Completion 2014-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
circulating tumor cells in blood | every 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of GI Oncology, Peking University Cancer Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li Y, Peng Z, Zhang X, Gong J, Shen L. [Value of serum human epithelial growth factor receptor 2 extracellular domain and circulating tumor cells in evaluating therapeutic response in advanced gastric cancer]. Zhonghua Wei Chang Wai Ke Za Zhi. 2017 Nov 25;20(11):1293-1299. Chinese. PMID 29178102